CLINICAL TRIAL: NCT02133820
Title: A 4-part, Single-dose, Open-label, Randomised, Crossover, Exploratory Study in Healthy Subjects to Assess the Influence of an Opioid Antagonist on How the Body Processes a Strong Painkiller, When Co-administered in a Fasted and Fed State.
Brief Title: A Study to Assess How the Body Processes a Strong Painkiller When it is Given Alongside a Drug That Counteracts the Side Effects of Strong Painkillers in a Fasted and Fed State.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mundipharma Research Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: HMX1507; 2013-005522-35 (EudraCT Number)
Record Dates: First submitted 2014-02-25; First posted 2014-05-08 (Estimated); Last update posted 2014-06-27 (Estimated); Status verified 2014-06

CONDITIONS: Pain
Keywords: Healthy Volunteer; Pharmacokinetics
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 12 hourly capsule fasted (Active Comparator): 4 mg 12 hourly capsule - strong pain killer fasted
  Interventions: Drug: 4 mg 12 hourly capsule - strong pain killer fed
- 12 hourly capsule fed (Active Comparator): 4 mg 12 hourly capsule - strong pain killer fed
  Interventions: Drug: 4 mg 12 hourly capsule - strong pain killer fasted
- 12 hourly capsule with antagonist fasted (Experimental): 4 mg 12 hourly capsule strong painkiller with antagonist fasted
  Interventions: Drug: 4 mg 12 hourly capsule strong painkiller with antagonist fed
- 12 hourly capsule with antagonist fed (Experimental): 4 mg 12 hourly capsule strong painkiller with antagonist fed
  Interventions: Drug: 12 hourly capsule strong painkiller with antagonist fasted)

INTERVENTIONS:
Drug: 4 mg 12 hourly capsule - strong pain killer fasted
  Other Names: MR2XXX
  Arms: 12 hourly capsule fed
Drug: 4 mg 12 hourly capsule - strong pain killer fed
  Other Names: MR2XXX
  Arms: 12 hourly capsule fasted
Drug: 12 hourly capsule strong painkiller with antagonist fasted)
  Other Names: MR2XXX
  Arms: 12 hourly capsule with antagonist fed
Drug: 4 mg 12 hourly capsule strong painkiller with antagonist fed
  Other Names: MR2XXX
  Arms: 12 hourly capsule with antagonist fasted

SUMMARY:
To assess whether an opioid antagonist has any impact on the release of a strong painkiller in the blood when it is given to healthy volunteers when they have eaten and also when they have fasted.

DETAILED DESCRIPTION:
This is an exploratory study to assess the influence of an opioid antagonist on the pharmacokinetics of a strong painkiller when co-administered in a fasted and fed state.

Determination is by measurement of drug concentrations in the blood at serial collection time points pre-dose until 32 hours post-dose, following an administration of a single oral dose. Pharmacokinetics parameters of AUC and Cmax are the primary endpoints.

ELIGIBILITY:
Healthy male or female subjects aged 18 to 55 inclusive Healthy and free of significant abnormal findings as determined by medical history, physical examination, vital signs, laboratory tests and ECG.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2014-04; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics parameters AUC and Cmax | Up to 32 hours

SECONDARY OUTCOMES:
Adverse Events | 7 to 10 days
  AEs will be recorded through spontaneous reporting
Vital Signs | 0 to 32 hours
  Vital signs - blood pressure, pulse rate, tympanic temperature and respiration rate
Clinical Laboratory Tests | Day 0 and Day 7-10
  Clinical laboratory tests - blood samples will be taken at screening and post-study medical for routine laboratory analysis (haematology, blood chemistry and urinalysis
ECG | Screening, 1 our post-dose and Day 7-10
  ECGs

CONTACTS AND LOCATIONS:
Locations (1):
- Quotient Clinical Limited, Nottingham, Nottinghamshire, United Kingdom